CLINICAL TRIAL: NCT02789956
Title: Clinical Outcomes of Implant- Versus Abutment-level Connection in Screw-retained Fixed Dental Prostheses
Brief Title: Internal vs. External Connection in Screw-retained Multi-units Bridges With Cad/Cam Milled Co/Cr Framework (ISUS-Atlantis)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute Franci (Other)
Responsible Party: Principal Investigator, Toia Marco, dr, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIS-14-083
Record Dates: First submitted 2016-05-29; First posted 2016-06-03 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Rehabilitation of Edentulous Area With an Implant Level Set-up
Keywords: Internal connection; Cobalt/Chrome; Cad-cam Framework; marginal bone level

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test: internal connection (Experimental): Evaluate marginal bone level (MBL) changes at implants that are placed semi-edentulous patient when they are treated with implant level Co/cr Cad/Cam framework.
  Interventions: Device: Internal vs. external cad cam co/cr framework
- Test: external connection (Active Comparator): Evaluate marginal bone level (MBL) changes at implants that are placed semi-edentulous patient when they are treated with abutment level Co/cr Cad/Cam framework.
  Interventions: Device: Internal vs. external cad cam co/cr framework

INTERVENTIONS:
Device: Internal vs. external cad cam co/cr framework
  Other Names: Astratech EV system, Dentsply HI

SUMMARY:
The aim of this study is to evaluate:

Primary objective The primary objective of the present study is to evaluate the marginal bone level changes when partially edentulous patients, treated with implants, received a multiunits screw retained fixed dental prosthesis with a Co/Cr milled framework with an Internal or External connection.

Secondary objective

1. Overall survival rate.
2. Soft tissue status by assessment of bleeding on probing (BoP) and probing pocket depth (PPD) at baseline and after 1,3,5 years.
3. Prosthetic survival rates including screw or abutment loosening, framework or veneer fractures.

DETAILED DESCRIPTION:
A randomized pilot study is designed to determine marginal bone changes between patients treated with a milled framework in Co/Cr if the connection is Internal or External for the rehabilitation of a partially edentulous area with a multiunit screw retained bridge. The investigation will be performed in one clinical centre affiliated to the Department of oral and maxillofacial surgery, Faculty of Odontology, Malmö University . In this center the clinician and the examiner will be the same person.

Following a screening examination, subjects who will meet the inclusion criteria, will sign the Informed Consent and will be enrolled in the study. The period of patient enrollment will begin on October 1st 2015 and ends September 31st 2016.

The patients will be randomized with a method based on the use of sealed opaque envelopes. The cases will be assigned to two different treatment groups:

Group A- Co/Cr milled framework with internal connection (Test) Group B- Co/Cr milled framework with external connection (Control)

-Pre-treatment Patient data, medical history, clinical and radiographic examination will be recorded for each patient. Clinical photographs will be taken in frontal, occlusal and lateral projections Periodontal, endodontic and open caries lesions will be treated prior to implant installation. All patients will receive careful oral hygiene instructions and training in self-performed plaque control measure.

Orthopantomogram at constant magnification and CT scan computed exams will be carried out.

Plaster models and diagnostic wax-up will be carried out.

-First Surgical Phase (Implant Installation) The patient will receive antibiotic prophylaxis (Amoxicillin 1gr) one hour prior to surgery and after the completion of implant installation until suture removal with 1gr three times a day. (If the patient is allergic to amoxicillin the examiner prescribes antibiotics at his own discretion at the same posology).

The surgical treatment will be performed under local anaesthesia. In case of remaining teeth, they will be extracted with conventional technique before implants' placement.

Implants will be placed according to the guidelines described in the Astra Tech Osseospeed EV® manual "Surgical procedures", using a two-stage protocol.

Implant spinning during the positioning of the cover screw will be registered as positive, if present, or negative.

The operation will be finalized by a careful adaption of the flaps by means of an accurate suture in order to obtain a full periosteal coverage.

Intraoral clinical photographs before, during and after surgery will be taken. -Post-operative care The patients will be instructed to rinse with chlorhexidine 0.12% mouthrinse and will be told to rinse with the antiseptic solution three times a day for 2 weeks. The patients will be advised to take NSAIDs for pain relief at their own discretion.

Liquid and semisolid food will be prescribed for the first post-operative week, after which the sutures will be removed.

Two weeks after the operation the denture will be properly relined until the second stage surgery.

Patients will be controlled at third and sixth weeks.

-Prosthetic procedures After eight weeks (+ 2) of implants healing a second stage surgery will be applied and Healing Abutment will be performed groups A while a Uni Abutment 33° connection procedure will be performed. In group B.

Impression with a customized spoon and Impregum material will be taken after one week from the second surgery and prosthetic procedure will be performed according to the Atlantis-Isus Dentsply Astra-tech prosthetic manual recommendations.

After 6 weeks (+ 2) from impression the definitive fixed dental prostheses screw retained multiunits bridge will be applied.

The prosthesis will be made to accomplish the normal hygienic procedures. All prosthetic procedures will be made in accordance to the Astra Tech procedures & products manuals.

The length of bridge cantilevers will be duly calculated to minimize implant overloading according to the Atlantis-Isus recommendations for both group.

-Post-prosthetic measurements Clinical measurements Clinical examinations will be performed immediately following the installation of the definitive prosthesis (Baseline-Loading) and after 1, 3, and 5 years. In particular, plaque and soft-tissue inflammation will be registered. Clinical photographs will be taken at each interval point.

Plaque: the presence of plaque will be scored at each implant site as well as at level of the remaining teeth on four surfaces (buccal, lingual/palatal, mesial, distal). The mean percentage of plaque harboring surfaces will be calculated using the case as the unit.

Soft-tissue inflammation: the presence of soft-tissue inflammation (bleeding on probing) will be assessed on buccal, lingual/palatal, mesial, distal aspects of each implant. The mean percentage of inflamed sites will be calculated using the case as the unit.

- Radiographic measurements

Peri-apical radiographs will be taken at prosthesis insertion (Baseline) and after 1, 3, and 5 years.

The radiographs will be taken with an X-ray apparatus supplied with a long cone by the examiner each visiting time. Rinn centrators will be used to ensure reproducibility in the measurement of marginal bone level change.

The radiographic images will be analysed at the Department of Radiology of Sahlgrenska Academy, Gothenburg University by experienced radiologists who will be otherwise not involved in the study.

9. STATISTICAL ANALYSIS

Results will be presented by appropriate descriptive and inferential statistic. Demographic and other baseline characteristics will be presented by means of descriptive statistics. Continuous variables will be presented by means of number of observations (N), minimum (min), median, maximum (max), mean and standard deviation (std). Discrete variables will be presented by frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Willingness to comply with all study requirements and to sign the IC.
* Systemic health.
* Compliance with good oral hygiene.
* Patients with at least 2 teeth to replace in any side of the jaws.

Exclusion Criteria:

* Patients treated with implant with bone defects associated with severe knife-edge ridges.
* Patients treated with bone defects resulting from tumor resection.
* Tobacco abuse (> 10 cigarettes/day).
* Severe renal and liver disease.
* History of radiotherapy in the head and neck region.
* Chemotherapy for treatment of malignant tumors at the time of the surgical procedure.
* Uncontrolled diabetes.
* Active periodontal disease involving the residual opposite dentition.
* Mucosal disease, such as lichen planus, in the areas to be treated.
* Poor oral hygiene.
* Non-compliant patients.
* Situations judged inconvenient(by the investigator) for the surgical treatment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2024-09 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Marginal bone resorption in millimeter from the implant to the bone crest. | 1 year
Marginal bone resorption in millimeter from the implant to the bone crest. | 3 year
Marginal bone resorption in millimeter from the implant to the bone crest. | 5 year

SECONDARY OUTCOMES:
Fracture of the prosthetic components | 1 year
Fracture of the prosthetic components | 3 year
Fracture of the prosthetic components | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Studiotoia Srl, Busto Arsizio, Varese, Italy